CLINICAL TRIAL: NCT00721279
Title: Sifrol Onset of Action and Impact: a 12-weeks Observational Study in Patients With Primary RLS
Brief Title: Sifrol (Pramipexole) Onset of Action and Impact: a 12-weeks Observational Study in Patients With Primary Restless Legs Syndrome
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.655
Record Dates: First submitted 2008-07-23; First posted 2008-07-24 (Estimated); Results first posted 2010-01-08 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Sifrol® (pramipexole dihydrochloride)

SUMMARY:
The objectives of the Post Market Surveillance (PMS) study are to evaluate the treatment effect of pramipexole on Restless Legs Syndrome (RLS) severity as measured by International Restless Legs Rating Scale and Global Clinical Impression - Improvement, to evaluate the time to reaching maintenance dose of pramipexole

ELIGIBILITY:
Inclusion Criteria:

* Primary Restless Legs Syndrome (i.e. idiopathic RLS)
* Indication for treatment with pramipexole
* Male or female patients older than 18 years

Exclusion Criteria:

* Any contraindications according to the Summary of Product Characteristics (SPC): hypersensitivity to pramipexole or to any of the excipients
* Current treatment with pramipexole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic RLS
Sampling Method: Non-Probability Sample
Enrollment: 549 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (127):
- Austria (127):
  - Boehringer Ingelheim Investigational Site, Absam
  - Boehringer Ingelheim Investigational Site, Absdorf
  - Boehringer Ingelheim Investigational Site, Afritz
  - Boehringer Ingelheim Investigational Site, Alkoven
  - Boehringer Ingelheim Investigational Site, Altenmarkt/Zauchensee
  - Boehringer Ingelheim Investigational Site, Anif
  - Boehringer Ingelheim Investigational Site, Au
  - Boehringer Ingelheim Investigational Site, Bad Goisern am Hallstättersee
  - Boehringer Ingelheim Investigational Site, Bad Schallerbach
  - Boehringer Ingelheim Investigational Site, Bad Vöslau
  - Boehringer Ingelheim Investigational Site, Baden
  - Boehringer Ingelheim Investigational Site, Bärnbach
  - Boehringer Ingelheim Investigational Site, Bleiburg
  - Boehringer Ingelheim Investigational Site, Bludenz
  - Boehringer Ingelheim Investigational Site, Bregenz
  - Boehringer Ingelheim Investigational Site, Bruck A.d. Mur
  - Boehringer Ingelheim Investigational Site, Deutschkreutz
  - Boehringer Ingelheim Investigational Site, Deutschlandsberg
  - Boehringer Ingelheim Investigational Site, Dornbirn
  - Boehringer Ingelheim Investigational Site, Ebensee
  - Boehringer Ingelheim Investigational Site, Faak am See
  - Boehringer Ingelheim Investigational Site, Ferlach
  - Boehringer Ingelheim Investigational Site, Fieberbrunn
  - Boehringer Ingelheim Investigational Site, Filzmoos
  - Boehringer Ingelheim Investigational Site, Fischamend
  - Boehringer Ingelheim Investigational Site, Fohnsdorf
  - Boehringer Ingelheim Investigational Site, Fritzens
  - Boehringer Ingelheim Investigational Site, Gallizien
  - Boehringer Ingelheim Investigational Site, Gallspach
  - Boehringer Ingelheim Investigational Site, Gaspoldshofen
  - Boehringer Ingelheim Investigational Site, Gerasdorf bei Wien
  - Boehringer Ingelheim Investigational Site, Gloggnitz
  - Boehringer Ingelheim Investigational Site, Gmunden
  - Boehringer Ingelheim Investigational Site, Grafenstein
  - Boehringer Ingelheim Investigational Site, Graz
  - Boehringer Ingelheim Investigational Site, Großklein
  - Boehringer Ingelheim Investigational Site, Grünbach
  - Boehringer Ingelheim Investigational Site, Haid
  - Boehringer Ingelheim Investigational Site, Halbturn
  - Boehringer Ingelheim Investigational Site, Hall in Tirol
  - Boehringer Ingelheim Investigational Site, Hart
  - Boehringer Ingelheim Investigational Site, Heidenreichstein
  - Boehringer Ingelheim Investigational Site, Hornstein
  - Boehringer Ingelheim Investigational Site, Innsbruck
  - Boehringer Ingelheim Investigational Site, Jenbach
  - Boehringer Ingelheim Investigational Site, Judenburg
  - Boehringer Ingelheim Investigational Site, Kapfenberg
  - Boehringer Ingelheim Investigational Site, Kematen
  - Boehringer Ingelheim Investigational Site, Klagenfurt
  - Boehringer Ingelheim Investigational Site, Kleinzell
  - Boehringer Ingelheim Investigational Site, Klosterneuburg
  - Boehringer Ingelheim Investigational Site, Krems
  - Boehringer Ingelheim Investigational Site, Kufstein
  - Boehringer Ingelheim Investigational Site, Laakirchen
  - Boehringer Ingelheim Investigational Site, Langenwang
  - Boehringer Ingelheim Investigational Site, Lavamünd
  - Boehringer Ingelheim Investigational Site, Längenfeld
  - Boehringer Ingelheim Investigational Site, Leibnitz, Styria
  - Boehringer Ingelheim Investigational Site, Leoben
  - Boehringer Ingelheim Investigational Site, Leopoldsdorf
  - Boehringer Ingelheim Investigational Site, Linz
  - Boehringer Ingelheim Investigational Site, Litschau
  - Boehringer Ingelheim Investigational Site, Litzelsdorf
  - Boehringer Ingelheim Investigational Site, Lofer
  - Boehringer Ingelheim Investigational Site, Marbach
  - Boehringer Ingelheim Investigational Site, Mattersburg
  - Boehringer Ingelheim Investigational Site, Meiningen
  - Boehringer Ingelheim Investigational Site, Melk
  - Boehringer Ingelheim Investigational Site, Micheldorf
  - Boehringer Ingelheim Investigational Site, Michelhausen
  - Boehringer Ingelheim Investigational Site, Mödling
  - Boehringer Ingelheim Investigational Site, Münzbach
  - Boehringer Ingelheim Investigational Site, Neufelden
  - Boehringer Ingelheim Investigational Site, Neunkirchen
  - Boehringer Ingelheim Investigational Site, Ottenheim
  - Boehringer Ingelheim Investigational Site, Pabneukirchen
  - Boehringer Ingelheim Investigational Site, Parndorf
  - Boehringer Ingelheim Investigational Site, Passail
  - Boehringer Ingelheim Investigational Site, Pernegg
  - Boehringer Ingelheim Investigational Site, Pinggau
  - Boehringer Ingelheim Investigational Site, Pischelsdorf
  - Boehringer Ingelheim Investigational Site, Poysdorf
  - Boehringer Ingelheim Investigational Site, Reichental
  - Boehringer Ingelheim Investigational Site, Ried im Innkreis
  - Boehringer Ingelheim Investigational Site, Roppen
  - Boehringer Ingelheim Investigational Site, Rüstorf
  - Boehringer Ingelheim Investigational Site, Saint Andrä
  - Boehringer Ingelheim Investigational Site, Saint Peter
  - Boehringer Ingelheim Investigational Site, Salzburg
  - Boehringer Ingelheim Investigational Site, Sandl
  - Boehringer Ingelheim Investigational Site, Sankt Florian
  - Boehringer Ingelheim Investigational Site, Sankt Gertraud
  - Boehringer Ingelheim Investigational Site, Sankt Pölten
  - Boehringer Ingelheim Investigational Site, Sankt Valentin
  - Boehringer Ingelheim Investigational Site, Sankt Veit an der Glan
  - Boehringer Ingelheim Investigational Site, Satteins
  - Boehringer Ingelheim Investigational Site, Schattendorf
  - Boehringer Ingelheim Investigational Site, Schörfling
  - Boehringer Ingelheim Investigational Site, Schwaz
  - Boehringer Ingelheim Investigational Site, Schwechat
  - Boehringer Ingelheim Investigational Site, Soielberg
  - Boehringer Ingelheim Investigational Site, Spielberg
  - Boehringer Ingelheim Investigational Site, Steinbrunn
  - Boehringer Ingelheim Investigational Site, Stockerau
  - Boehringer Ingelheim Investigational Site, Strallegg
  - Boehringer Ingelheim Investigational Site, Telfs
  - Boehringer Ingelheim Investigational Site, Veitsch
  - Boehringer Ingelheim Investigational Site, Vienna
  - Boehringer Ingelheim Investigational Site, Villach
  - Boehringer Ingelheim Investigational Site, Vorchdorf
  - Boehringer Ingelheim Investigational Site, Völs
  - Boehringer Ingelheim Investigational Site, Wagna
  - Boehringer Ingelheim Investigational Site, Walding
  - Boehringer Ingelheim Investigational Site, Wals
  - Boehringer Ingelheim Investigational Site, Wartberg
  - Boehringer Ingelheim Investigational Site, Wattens
  - Boehringer Ingelheim Investigational Site, Weer
  - Boehringer Ingelheim Investigational Site, Weiz
  - Boehringer Ingelheim Investigational Site, Weißkirchen in Steiermark
  - Boehringer Ingelheim Investigational Site, Wels
  - Boehringer Ingelheim Investigational Site, Wiener Neudorf
  - Boehringer Ingelheim Investigational Site, Wiener Neustadt
  - Boehringer Ingelheim Investigational Site, Wieselburg
  - Boehringer Ingelheim Investigational Site, Wilhelmsburg
  - Boehringer Ingelheim Investigational Site, Windhaag
  - Boehringer Ingelheim Investigational Site, Wolkersdorf
  - Boehringer Ingelheim Investigational Site, Zirl

RESULTS

PARTICIPANT FLOW:
Groups:
- De-novo Patients: Patients that had not been treated for RLS at baseline
- Pre-treated Patients: Patients that had been treated for RLS at baseline
Period: Overall Study
Arm/Group | De-novo Patients | Pre-treated Patients
Started | 452 | 97
Completed | 416 | 73
Not Completed | 36 | 24
Not completed — Lack of Efficacy | 6 | 3
Not completed — Tolerability insufficient | 5 | 2
Not completed — Withdrawal by Subject | 13 | 3
Not completed — Other | 12 | 16

BASELINE CHARACTERISTICS:
Population: SAF - Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | De-novo Patients | Pre-treated Patients | Total
Number analyzed (Participants) | 452 | 97 | 549
Age, Continuous [Mean (Standard Deviation); unit: years] — N= 432 - De-novo, 85 - Pre-treated, 517- Total
  years | 66.48 (12.87) | 67.81 (12.61) | 66.69 (12.82)
Sex/Gender, Customized [Number; unit: participants]
  Female | 317 | 66 | 383
  Male | 131 | 23 | 154
  missing | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Frequency Analysis for Baseline Pattern of RLS Symptoms
Description: Severity of RLS was rated using the International RLS Severity Scale. This scale measures the severity of RLS symptoms and comprises of 10 questions with 5 possible answers, each answer scored from 0-4 points and is classified into 5 RLS severity groups: 0 points = no symptoms, 1-10 points = mild, 11-20 points = moderate, 21-30 points = severe, 31-40 points = very severe.
Time Frame: Baseline
Population: Full analysis set (FAS)
Measure: Number; unit: percentage of participants
Arm/Group | De-novo Patients | Pre-treated Patients
Number analyzed (Participants) | 440 | 83
percentage of participants
  Mild | 0.7 | 2.4
  Moderate | 19.3 | 18.1
  Severe | 62.0 | 55.4
  Very Severe | 18.0 | 24.1

2. Primary Outcome: Change in Total Scores of IRLS (International Restless Legs Rating Scale)
Description: The International Restless Legs Syndrome Rating Scale (IRLS) is a rating scale used to assess the severity of RLS symptoms. The IRLS consists of 10 items, each of which is rated from 0 to 4 points, higher values denoting an increased severity of symptoms. Maximum total score is 40. Score totals are grouped into four levels of severity: 1-10 points = mild RLS, 11-20 points = moderate RLS, 21-30 points = severe RLS, and 31-40 = very severe RLS.
  The change from baseline was calculated as baseline minus the week 12 value.
Time Frame: Baseline and final visit (week12)
Population: Only those patients of the full analysis set with an evaluation of the IRLS at visit 3 were included
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | De-novo Patients | Pre-treated Patients
Number analyzed (Participants) | 428 | 80
scores on a scale | 17 [13.00 to 22.00] | 16 [11.00 to 22.75]

3. Primary Outcome: Change in Global Clinical Impression - Improvement (CGI-I) Scale
Description: The Clinical Global Impression Improvement scale (CGI-I) requires the clinician to rate how much the patient's illness has improved or worsened relative to a baseline state. A patient's illness is compared to change over time and rated as: very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse
Time Frame: baseline and final visit (week 12)
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | De-novo Patients | Pre-treated Patients
Number analyzed (Participants) | 440 | 83
percentage of participants
  Very much improved | 47.0 | 44.6
  Much improved | 45.5 | 42.2
  Minimally improved | 3.0 | 8.4
  No change | 1.8 | 2.4
  Minimally worse | 0.0 | 0.0
  Much worse | 0.2 | 0.0
  Very much worse | 0.0 | 0.0
  missing | 2.5 | 2.4

4. Primary Outcome: Frequency of Adverse Events
Description: Frequency of patients with any adverse event, causally related adverse events and serious adverse events
Time Frame: Up to 16 weeks
Population: Safety Analysis Set (SAF)
Measure: Number; unit: participants
Groups:
- Overall: All Patients
Arm/Group | Overall
Number analyzed (Participants) | 549
participants
  Any adverse event | 25
  Causally related adverse event | 7
  serious adverse events | 2

5. Primary Outcome: Correlation of the Change in IRLS at End of Titration and at Final Visit
Description: Correlation of the change in IRLS at end of titration and at final visit
Time Frame: Up to 12 weeks
Population: Full Analysis Set (FAS)
Measure: Number; unit: percentage of patients
Arm/Group | Overall
Number analyzed (Participants) | 523
percentage of patients
  End of titration - Deterioration (n=517) | 0.0
  End of titration - No change (n=517) | 19.7
  End of titration - Improvement (n=517) | 80.3
  Final Visit - Deterioration | 0.2
  Final Visit - No change | 5.4
  Final Visit - Improvement | 94.5

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: The Safety Analysis Set (SAF) including the data of all 549 patients reported to have received at least one dose of pramipexole.
Arm/Group | De-novo Patients | Pre-treated Patients
Serious Adverse Events (participants affected / at risk) | 0/452 | 2/97
Other Adverse Events (participants affected / at risk) | 0/452 | 0/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | De-novo Patients (N=452) | Pre-treated Patients (N=97)
Epilepsy (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Suicidal Tendency (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.